CLINICAL TRIAL: NCT06060613
Title: A Phase 1/2, Open-Label Study to Investigate the Safety and Efficacy of Membrane Bound IL15 Expressing Tumor-Infiltrating Lymphocytes (OBX-115) In Participants With Advanced Solid Tumors
Brief Title: Safety and Efficacy of OBX-115 in Advanced Solid Tumors
Acronym: Agni-01
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Obsidian Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: OBX115-23-01
Record Dates: First submitted 2023-09-22; First posted 2023-09-29 (Actual); Last update posted 2025-08-29 (Actual); Status verified 2025-07

CONDITIONS: Tumor Skin; Metastatic Melanoma; Melanoma; Lung Cancer; Metastatic Lung Cancer; Non Small Cell Lung Cancer; Metastatic Non Small Cell Lung Cancer
Keywords: Adoptive cell therapy; Tumor Infiltrating Lymphocytes; TIL; Melanoma; Lung Cancer
MeSH Terms: conditions — Skin Neoplasms; Melanoma; Lung Neoplasms; Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Intervention Model Description: Single group assignment
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Participants with advanced solid tumors (Experimental): Participants will receive conditioning therapy prior to administration of OBX-115 regimen.
  Interventions: Biological: OBX-115

INTERVENTIONS:
Biological: OBX-115 — A tumor sample is obtained from each participant for autologous OBX-115 manufacture.
  After lymphodepletion including cyclophosphamide and fludarabine, participant will receive OBX-115 infusion, followed by short courses of acetazolamide.

SUMMARY:
This is a study to investigate the safety and efficacy of an investigational OBX-115 regimen in adult participants with advanced solid tumors.

DETAILED DESCRIPTION:
Primary Objective (Phase 1):

• Assess the safety and tolerability of OBX-115 regimen

Primary Objective (Phase 2):

• Evaluate preliminary efficacy of OBX-115 regimen as measured by the investigator using objective response rate (ORR) per Response Evaluation Criteria in Solid Tumors (RECIST) v1.1

Secondary (Phase 1):

• Assess preliminary efficacy of OBX-115 regimen by evaluating ORR

Secondary (Phase 2):

• Evaluate safety and tolerability of OBX 115 based on the collected AE data

Secondary (both Phase 1 and Phase 2):

* Evaluate duration of response (DOR): To evaluate the duration from the time that criteria are met for CR or PR per RECIST v1.1 as assessed by the investigator until disease progression or death due to cancer.
* Evaluate disease control rate (DCR): To evaluate the percentage of participants with a best overall confirmed response of CR or PR at any time plus stable disease (SD) for at least 4 weeks per RECIST v1.1 as assessed by the investigator.
* Evaluate progression-free survival (PFS): To evaluate the time from the date of OBX-115 infusion until disease progression per RECIST v1.1 as assessed by the investigator or death due to any cause.
* Evaluate overall survival (OS): To evaluate the time from the date of OBX-115 infusion to death due to any cause
* Evaluate feasibility of the manufacturing process: Evaluated as the proportion of OBX-115 products initiated for manufacturing that pass release criteria for infusion.

ELIGIBILITY:
Inclusion Criteria:

1. Participant must be 18 years of age or older at the time of signing the informed consent.
2. Participant has a histologically confirmed diagnosis of advanced/metastatic melanoma ore relapsed refractory metastatic non-small cell lung cancer (NSCLC).
3. Melanoma participant experienced documented radiographic disease progression after systemic therapy containing a programmed cell death protein 1 (PD-1)/programmed death ligand 1 (PD-L1) blocking antibody. Participants with melanoma must not exceed 2 prior lines of systemic therapy. Neoadjuvant/Adjuvant treatment will not be considered a prior line of systemic therapy unless the participant progressed during or within the 12 weeks after the last dose of the adjuvant PD-1/PD-L1 blocking antibody. Participants with non-small cell lung cancer should have relapsed or are refractory to approved systemic therapies (approved ICI-based regimen for all appropriate participants and/or an approved targeted therapy for known molecular abnormalities if applicable to their disease). Participant must not have been exposed to both taxane and gemcitabine.
4. Participant is assessed as having at least one lesion (or aggregate lesions) suitable for OBX-115 generation.
5. After tumor tissue procurement, the participant will have at least one remaining measurable lesion, as defined by RECIST v1.1.
6. Participant has an Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1 and an estimated life expectancy of greater than 6 months.
7. Participant has recovered from all prior anticancer treatment-related AEs to at least Grade 1 (per Common Terminology Criteria for Adverse Events [CTCAE]).
8. Participants must have completed post-operative recovery from any prior surgical procedures with wound healing and resolution of all surgical complications prior to planned tumor procurement surgery.
9. Both male and female (women of childbearing potential) participants agree to the follow protocol specified contraceptive and/or abstinence requirements.
10. Participant has protocol specified hematologic parameters for absolute neutrophil count (ANC) and platelet count.
11. Participant has adequate cardiac, liver, lung, and kidney organ function as specified in the protocol.

Exclusion Criteria:

1. Participant has melanoma of uveal origin or its other genetic equivalents (e.g. GNA11 and GNAQ).
2. Participant has a history of brain metastases or leptomeningeal disease. Participants may be considered for enrollment if they have 4 or fewer brain metastatic lesions that are up to 1.5cm in diameter that have been treated, if clinically indicated.
3. Participant has an active medical illness(es) that, in the opinion of the Investigator, would pose increased risks for study participation.
4. Participants with non-small cell lung cancer with refractory and clinically significant pleural effusions.
5. Participant has any form of primary or acquired immunodeficiency.
6. Participant has a history of hypersensitivity to any component of the study intervention.
7. Participant had another primary malignancy within the previous 3 years (with protocol specified exceptions).
8. Participant has a history of allogeneic organ transplant, allogeneic cell therapy, or genetically engineered cell therapy. Prior engineered TIL cell therapy is allowed.
9. Participant requires systemic steroid therapy of greater than10 mg/day of prednisone or equivalent.
10. Participant received a live or attenuated vaccination within 28 days prior to the start of lymphodepletion (LD).
11. Participant has evidence of positive infectious disease screening and/or any active uncontrolled viral, bacterial, or fungal disease requiring ongoing systemic treatment or identified during screening.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Estimated)
Dates: Start 2023-10-25 (Actual); Primary Completion 2028-06-30 (Estimated); Study Completion 2028-06-30 (Estimated)

PRIMARY OUTCOMES:
Incidence and nature of dose-limiting toxicities (DLTs) | 28 Days
  • Incidence of dose-limiting toxicities (DLTs) during the first 28 days after OBX-115 infusion (Phase 1).
The proportion of participants who have a confirmed complete response (CR) or partial response (PR) per RECIST v1.1 | 2 years
  • The proportion of participants who have a confirmed complete response (CR) or partial response (PR) per RECIST v1.1 as assessed by the Investigator from the date of OBX-115 infusion until disease progression, death, start of a new anticancer therapy, withdrawal of consent, or end of study, whichever comes first (Phase 2)

SECONDARY OUTCOMES:
The proportion of participants who have a confirmed CR or PR per RECIST v1.1 | 2 years
  • The proportion of participants who have a confirmed CR or PR per RECIST v1.1 as assessed by the Investigator from the date of OBX-115 infusion until disease progression, death, start of a new anticancer therapy, withdrawal of consent, or end of study, whichever comes first (Phase 1)
Incidence of AEs | 2 years
  • Incidence of treatment-emergent adverse events (TEAEs), including SAEs, study intervention related AEs, and AEs leading to early discontinuation of study intervention or withdrawal from the Assessment Period or death up to 2 years after initiation of study intervention

CONTACTS AND LOCATIONS:
Locations (9):
- United States (9):
  - The Angeles Clinic and Research Institute (Melanoma), Los Angeles, California
  - USC Norris Comprehensive Cancer Center (Melanoma/NSCLC), Los Angeles, California
  - Stanford Cancer Institute (Melanoma/NSCLC), Stanford, California
  - Orlando Health Cancer Institute (Melanoma/NSCLC), Orlando, Florida
  - James Graham Brown Cancer Center (Melanoma/NSCLC), Louisville, Kentucky
  - Memorial Sloan Kettering (Melanoma/NSCLC), New York, New York
  - The Ohio State University, Columbus, Ohio
  - Allegheny Research Institute (Melanoma/NSCLC), Pittsburgh, Pennsylvania
  - M.D. Anderson Cancer Center (Melanoma/NSCLC), Houston, Texas

IPD SHARING:
Plan to Share IPD: No